CLINICAL TRIAL: NCT02833818
Title: Growth and Development of Premature Babies
Brief Title: Effect of Intensive Dietary Intervention in Children With Birth Weight Between 1500 and 2000 g
Acronym: CAKE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elin Wahl Blakstad (Other)
Responsible Party: Sponsor-Investigator, Elin Wahl Blakstad, dr. Elin Wahl Blakstad, University Hospital, Akershus
Organization: University Hospital, Akershus (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AkershusUH
Record Dates: First submitted 2016-01-11; First posted 2016-07-14 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Perinatal Disorders of Growth and Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAKE-intervention (Experimental): Increased nutrition and dietary consultations. Growth rate followed by clinical nutritionists that supply high protein and energy if growth rate deviates from 17g/kg/day
  Interventions: Dietary Supplement: CAKE-intervention
- CAKE-control (Active Comparator): nutrition according to established procedures in the neonatal intensive care unit (NICU)
  Interventions: Dietary Supplement: CAKE-control

INTERVENTIONS:
Dietary Supplement: CAKE-intervention — Increased protein and energy supplementation and conversations
  Other Names: clinical nutritionist, high protein and energy
  Arms: CAKE-intervention
Dietary Supplement: CAKE-control — nutrition according to established procedures
  Arms: CAKE-control

SUMMARY:
There are few scientific reports on preterm infants with birth weights between 1500 and 2000g. Adequate and properly balanced supply of nutrients believed to better growth and cognitive development in this patient group, and optimized nutrition is an important part of treatment There is a need for more studies that can provide knowledge of growth and weight development in preterm and small for gestational age (SGA) infants with a birth weight between 1500 and 2000g.

DETAILED DESCRIPTION:
There has been little focus, at least there are few scientific reports on preterm infants with birth weights between 1500 and 2000g, at least in Norway. Studies have shown the benefit of enhanced protein and energy supplements in very low birth weight infants (VLBW, birth weight < 1500g), regarding growth and neurodevelopment . Adequate and properly balanced supply of nutrients is believed to give better growth and cognitive development in premature infants with slightly higher birth weight, i.e between 1500 and 2000g (1). In an intervention study of VLBW children at four Norwegian hospitals we found lower supply of energy and protein than international recommendations (2). A larger proportion of premature children were stunted growth (weight below 10 percentile for age) during hospitalization. Although this applies to preterm infants with birth weight less than 1500 g, this may also be the case for larger premature patients.

More studies that can provide knowledge of growth rate, weight and neurodevelopmental outcomes in preterm and small for gestational age (SGA) infants are warranted. This study examines those with birth weight between 1500 and 2000g. Overall, this may provide new and useful knowledge that can help to optimize the nutrition to preterm and SGA infants with a this range of birth weights

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight between 1500 and 2000g.
2. No invasive catheters or ventilator (wish homogeneous group).
3. No malformations or chromosomal disorders.
4. Parents give informed written consent
5. Born at study hospitals

Exclusion Criteria:

1. Birth weight below 1500 and above 2000g.
2. Invasive catheters or ventilator.
3. Malformations or chromosomal disorders.

Ages: 26 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2010-10 (Actual); Primary Completion 2022-02-20 (Estimated); Study Completion 2022-02-20 (Estimated)

PRIMARY OUTCOMES:
Growth at 4 months corrected months age | From birth until 4 months postmenstrual age (PMA)
  Growth from birth, during hospital stay, at discharge/term and at 4 months PMA.
Breastfed, full or partly, and solid food at 4 months PMA | From birth until 4 months PMA
  Eating habits at discharge/term and at 4 months PMA .

CONTACTS AND LOCATIONS:
Overall Officials: Britt Nakstad, PhD MD, Study Director — Project leader

IPD SHARING:
Plan to Share IPD: Undecided